CLINICAL TRIAL: NCT02933983
Title: Study of the Microbiota and the Potential of Probiotics for Chronic Rhinosinusitis
Brief Title: Microbiota Upper Respiratory Tract
Acronym: ProCure
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, prof. dr. Olivier Vanderveken, MD, PhD, University Hospital, Antwerp
Other Study IDs: B300201524257
Record Dates: First submitted 2016-07-14; First posted 2016-10-14 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Microbiota Upper Respiratory Tract

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group (healthy): Participants who do not suffer from acute or chronic airway infections
  Interventions: Other: no intervention, compare URT microbiome healthy control group-chronic rhinosinusitis patients
- CRS patients: Patients who suffer from chronic rhinosinusitis
  Interventions: Other: no intervention, compare URT microbiome healthy control group-chronic rhinosinusitis patients

INTERVENTIONS:
Other: no intervention, compare URT microbiome healthy control group-chronic rhinosinusitis patients

SUMMARY:
The aim of this study is to investigate whether the microbiota in the upper respiratory tract (URT) (nose, nasopharynx and sinuses) of chronic rhinosinusitis (CRS) patients is disturbed compared to healthy individuals. Therefore, bacterial DNA from swabs, aspirates and tissue will be isolated via commercially available DNA extraction kits, followed by Illumina MiSeq sequencing in order to identify the bacterial species present in these samples. Special attention will go to microbial species that are overrepresented in the healthy populations as potential health promoting microbes (i.e. probiotics). A better understanding of the URT microbiome might help us to better understand the pathology of CRS and might help to develop new microbiota-based strategies for CRS.

ELIGIBILITY:
Exclusion Criteria healthy population:

* no use of antibiotics in the past year
* no acute or chronic airway infections
* no cancer
* no autoimmune diseases
* pregnant women

Exclusion Criteria CRS population:

--> no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population involves both healthy individuals and CRS patients.
Sampling Method: Non-Probability Sample
Enrollment: 325 (Actual)
Dates: Start 2015-05; Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
differences in bacterial communities colonizing the upper respiratory tract between healthy individuals and CRS patients measured via Illumina MiSeq | up to 4 years before all samples from both groups are collected and processed
  After Illumina MiSeq sequencing, bio-informatic tools will be used to cluster bacteria into operational taxonomic units (OTUs). Based on these OTUs, we will compare the composition of the bacteria in the sampled niches and compare this composition between healthy individuals and chronic rhinosinusitis patients. We will specifically screen for OTUs that are over- or underrepresented in both populations. Furthermore, special attention will go to screen for the typical nasopharyngeal pathogens such as Staphylococcus aureus, Streptococcus pneumoniae, Haemophilus influenzae, ... and also to beneficial microbes such as lactic acid bacteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Boeck I, Wittouck S, Martens K, Claes J, Jorissen M, Steelant B, van den Broek MFL, Seys SF, Hellings PW, Vanderveken OM, Lebeer S. Anterior Nares Diversity and Pathobionts Represent Sinus Microbiome in Chronic Rhinosinusitis. mSphere. 2019 Nov 27;4(6):e00532-19. doi: 10.1128/mSphere.00532-19. PMID 31776238